CLINICAL TRIAL: NCT03257306
Title: Magnetic Ureteral Stent Symptoms - a Comparison to Standard Ureteral Stent as Perceived By the Patient (MAGUSS)
Acronym: MAGUSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Kuopio University Hospital (Other); Satakunta Central Hospital (Other); Jyväskylä Central Hospital (Other)
Responsible Party: Principal Investigator, Kari Syvanen, Principal Investigator, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMTK 66/1801/2017
Record Dates: First submitted 2017-08-02; First posted 2017-08-22 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Urinary Tract Stone; Kidney Stone
Keywords: Urinary tract stone; ureter double-J stent
MeSH Terms: conditions — Urinary Calculi; Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Prospective randomized, single-blinded, multi-institutional, non-inferiority study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magnetic double-J ureteric stent (Active Comparator): Double-J ureteric stent removed using magnet
  Interventions: Procedure: ureteral double-J stent removal using magnet; Procedure: ureteral double-J stent removal using cystoscopy
- Standard double-J ureteric stent (Active Comparator): Double-J stent removed using cystoscopy
  Interventions: Procedure: ureteral double-J stent removal using magnet; Procedure: ureteral double-J stent removal using cystoscopy

INTERVENTIONS:
Procedure: ureteral double-J stent removal using magnet — Double-J ureteric stent removed using magnet
Procedure: ureteral double-J stent removal using cystoscopy — Double-J ureteric stent removed using cystoscopy

SUMMARY:
The specific aim of this study is to validate our hypothesis that the magnetic ureteral stents have the same amount of adverse effects as the more commonly used non-magnetic ureteral stents. If this hypothesis would be confirmed then the usage of magnetic ureteral stents would be justified for both reducing patient discomfort by way of fewer cystoscopies and possibly also decreasing the overall expenditures of treatment.

DETAILED DESCRIPTION:
Many urological procedures involving the kidney and the ureters require a stent replacement to avoid un-wanted adverse invents caused by the procedure itself. The stenting, however, predisposes the patient to adverse effects of its own and the application and removal of the stent is a notable monetary expense. The use of magnetic ureteral stents that can be removed via catheter instead of requiring an additional cystoscopy for removal would reduce the discomfort to patients and also possibly decrease the expenditures of the overall treatment. However, the comparability of standard ureteral stents and the magnetic ureteral stents is largely unknown due to there being no published research on the subject as of this time. The specific aim of this study is to validate our hypothesis that the magnetic ureteral stents have the same amount of adverse effects as the more commonly used non-magnetic ureteral stents.

The design is as prospective randomized, single-blinded, multi-institutional, non-inferiority study conducted in Hospital Districts of Southwest Finland, Päijät-Häme, Pohjois-Savo, Satakunta and Keski-Suomi. Using age and gender stratification, patients are randomised 1:1 fashion into having a magnetic (n=85) or standard ureter stent (n=85). The primary objectives are the mean differences between the two groups in pain and urinary symptoms scores determined by the Ureteral Stent Symptom Questionnaire (USSQ) 4 weeks after stent placement.

The patients will be recruited starting from the 4rd quarter of 2018 and ending during the 3rd quarter of 2020. Preliminary analysis of all results will be available in September 2020 and reports are expected to be written during December 2020.

ELIGIBILITY:
Inclusion Criteria:

* Language spoken: Finnish
* Clinically evaluated need for short term ureter stenting in course of extracorporeal shockwave lithotripsy-treatment or after pyeloscopy
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethics Committee (EC) approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* Current use of alpha blockers
* Patients undergoing emergency ureteroscopy and stenting
* Patients with a long term ureter stents
* Any other conditions that might compromise patients safety, based on the clinical judgment of the responsible urologist

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in Pain score in Ureteral Stent Symptom Questionnaire (USSQ) | 4 weeks after stent placement and 4 weeks after stent removal
  4 weeks after stent placement. [5] Less than 5 points of difference between the two study groups is considered as clinically insignificant.

SECONDARY OUTCOMES:
General health score in Ureteral Stent Symptom Questionnaire (USSQ) | 4 weeks after stent placement and 4 weeks after stent removal
  4 weeks after stent placement. Scores less than 4 points of difference between the two study groups is considered as clinically insignificant.
Sexual score in Ureteral Stent Symptom Questionnaire (USSQ) | 4 weeks after stent placement and 4 weeks after stent removal
  4 weeks after stent placement. Scores less than 4 points of difference between the two study groups is considered as clinically insignificant.
Working performance score in Ureteral Stent Symptom Questionnaire (USSQ) | 4 weeks after stent placement and 4 weeks after stent removal
  4 weeks after stent placement. Scores less than 4 points of difference between the two study groups is considered as clinically insignificant.
Urinary symptom score in Ureteral Stent Symptom Questionnaire (USSQ) | 4 weeks after stent placement and 4 weeks after stent removal
  4 weeks after stent placement. Scores less than 4 points of difference between the two study groups is considered as clinically insignificant.

OTHER OUTCOMES:
The discomfort experienced by the patients during stent removal determined in 100mm Visual Analogue Scale (VAS). | 4 weeks after stent placement
  More than 10mm difference between the two groups is considered as clinically significant.
The number of unsuccessful removals of the magnetic stent. | 4 weeks after stent placement
  Unsuccessful removal using magnet

CONTACTS AND LOCATIONS:
Overall Officials: Kari T Syvänen, MD, PhD, Principal Investigator — Turku University Hospital
Locations (3):
- Finland (3):
  - Keski-Suomi Central Hospital, Jyväskylä
  - Satakunta Central Hospital, Pori
  - Turku University Hospital, Turku